CLINICAL TRIAL: NCT01154257
Title: Comparison of Foam Swabs Versus Toothbrushes in Removing Dental Plaque From Orally Intubated Mechanically Ventilated Patients
Brief Title: Comparison of Swabs and Toothbrushes in Cleaning the Teeth of Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/MRE09/44
Record Dates: First submitted 2010-06-14; First posted 2010-06-30 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2020-01

CONDITIONS: Dental Plaque; Gingivitis
Keywords: Dental plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cleaning teeth with toothbrush (Experimental): Following randomisation one side of the mouth (split mouth study) will be assigned to cleaning teeth with a toothbrush
  Interventions: Procedure: Cleaning of teeth with a toothbrush
- Cleaning teeth with foam swab (Experimental): Following randomisation one side of the mouth (split mouth study) will be assigned to cleaning teeth with a faom swab
  Interventions: Procedure: Cleaning of teeth with a foam swab

INTERVENTIONS:
Procedure: Cleaning of teeth with a toothbrush — This is a split mouth study where patients will have one side of their mouth randomised for teeth cleaning with a toothbrush. Cleaning will be twice daily from recruitment until day seven.
  Arms: Cleaning teeth with toothbrush
Procedure: Cleaning of teeth with a foam swab — This is a split mouth study where patients will have one side of their mouth randomised for teeth cleaning with a foam swab. Cleaning will be twice daily from recruitment until day seven.
  Arms: Cleaning teeth with foam swab

SUMMARY:
Cleaning the mouth is difficult in critically ill patients who require support from a breathing machine (ventilator). This is because the plastic (endotracheal) tube which is a necessary interface between patient and ventilator impedes cleaning. New evidence suggests that poor oral health may be linked to ventilator associated pneumonia. Throughout the world both toothbrushes and foam swabs are used to clean the teeth and remove dental plaque, however it is unknown if one method is more effective than the other. The purpose of this study is to establish which (if any) method is most effective at removing plaque in this population of patients.

DETAILED DESCRIPTION:
Study Objective: The principle aim of this work is to determine whether foam swabs or toothbrushes offer the most effective method of removing dental plaque in orally intubated mechanically ventilated patients.

The secondary objective is to profile the microbiological flora in dental plaque, endotracheal tube and lung. In addition, collection of both plaque samples, used endotracheal tubes (ETTs) and non-directed bronchoalveolar lavage (NBL) will allow us to determine whether oral microorganisms contribute to biofilm formation within the ETT and potentially promote VAP. The findings of this study will not only enhance our knowledge on the organisms involved in promoting biofilms on ETT, but may also highlight potential management strategies to reduce their formation.

Study Population: Critically ill adult patients admitted to the intensive care unit at the University Hospital of Wales, Cardiff in whom mechanical ventilation has been initiated.

Recruitment: All patients satisfying inclusion and exclusion criteria, admitted to the adult ICU at the University Hospital of Wales from the start date of the study will be considered eligible for recruitment. Patients identified by the duty consultant will be notified to the research team. Consent will be obtained and in total 50 patients will be recruited.

Interventions: This is a split mouth design study whereby the intervention (cleaning with a foam swab or toothbrush) is performed on one side of the mouth. For example foam swab left side of mouth and toothbrush right side of mouth. Cleaning will be performed daily for a minimum of 24-hours or until extubation or up to seven days after recruitment, whichever is the shorter.

Non-directed bronchoalveolar lavages (NBLs) will be taken on a Monday and Thursday and when clinically indicated (for example a suspected VAP). This involves the insertion of a sterile suction catheter into the lung, 10-20ml of sterile saline is instilled and drawn back, and placed in a sterile universal. The sample will be split into two when there is a suspected infection, one half going to the UHW microbiology laboratory as usual, the other half will be profiled as part of the study. If there is no suspected infection all of the sample will be profiled as part of the study.

Methods: Following recruitment, patients will have their teeth cleaned twice a day with sterile water for 2 minutes using a 'baby toothbrush' and foam swab, the side to which the cleaning method is allocated will be randomised. One minute of cleaning assigned to each side of the mouth.

A modified Silness and Loe plaque score (Scannapieco et al 1992) and gingival index (Loe and Silness 1963) will be recorded prior to cleaning and then each morning following cleaning throughout the duration of the study. The plaque index will be recorded on the upper and lower first molars, first bicuspid and central incisors on each side of the mouth from the buccal surface. The plaque index score will be an average of the six teeth on each side. For patients with missing index teeth, the remaining teeth in closest proximity will be scored. The gingival index will be scored on the same teeth.

Following recording of the plaque and gingival index plaque samples will be collected on the same teeth as used for the plaque score. Samples of supragingival plaque will then be collected from the gingival third portion of the targeted teeth using a sterile curette prior to initiation of oral care and then once a day before cleaning. Plaque will immediately be inoculated into 1ml of microbiological transport medium. The transport medium will be diluted in a serial decimal manner in phosphate buffered saline prior to inoculation of agar plates using a spiral plating system (Don Whitley Scientific). The following agars will be used to culture the microorganisms: Blood Agar (aerobic bacteria), Fastidious Anaerobe Agar (anaerobic bacteria) and CHROMagar Candida (Candida and yeast species). Differential counts of lactose fermenting enteric bacteria will be through the use of MacConkey Agar, whilst Staphylococcus species (coagulase positive and coagulase negative) will be detected using Mannitol Salt Agar (MSA). The inoculated media will be incubated under appropriate gaseous environments at 37°C for 48 h (aerobes) or 7 d (anaerobes). A total aerobic microbial count from each side will be obtained from the blood agars and expressed as total colony forming units (CFUs).

Identification of each distinct colony morphotype will be through extensive phenotypic investigation. Tests will involve Gram staining, oxidase and catalase activity and biochemical profiling through a range of test systems. The biochemical test systems will include the APICoryne system (Gram-positive bacilli), APIStrep system (catalase-negative Gram-positive cocci), APIStaph and ID32Staph (catalase-positive Gram-positive cocci). Oxidase-negative, Gram-negative bacilli will be profiled using the API20E test whilst, oxidase-positive Gram-negative bacilli will be profiled using the API NE. Fungal organisms (Candida and yeast species) will be identified based on colony colour and appearance on the differential medium, CHROMagar and by biochemical profiling with the Auxocolour 2 system (biorad).

NBLs collected as outlined in the section on interventions above. Identification of the organisms present within the NBL samples will be done using the cultural methods outlined above.

If patients are extubated during the study then the endotracheal tube will be collected and transferred to the laboratory. Processing of ETT will involve dividing each tube into sections for either quantitative identification of organisms by microbial culture, molecular analysis or microscopical imaging.

Sections of each ETT will initially be placed in 2 ml of phosphate buffered saline and vortex mixed for 30 s with sterilised glass beads to disrupt biofilm aggregates. The PBS solution will then be removed and diluted serial decimally, 106-fold.

Identification of the organisms present within the biofilms will be done using the cultural methods outlined above, together with supplemental molecular analysis (outlined below).

16S ribosomal RNA gene-defined bacterial contamination of endotracheal tubes Sections from each region of recovered endotracheal tubes will be analysed using molecular procedures. The method will involve the extraction of total DNA from 500 µl of the specimens using a Puregeneâ bacterial DNA isolation kit (Gentra Systems). Universal bacterial primer pairs, d88 and e94 (Paster et al, 2001) and primers specific for target organisms (Porphyromonas gingivalis, Streptococcus mutans, Pseudomonas aeruginosa and Staphylococcus aureus) will then be used to amplify the 16S rRNA gene targets within the extracted samples using standard PCR and reaction conditions. Negative controls will include a reagent control (sterile water as PCR template) and a sample preparation control (sterile water used in place of the original sample and exposed to the entire extraction protocol). Positive controls of template DNA from known species of P. gingivalis, S. aureus and mutans will also be included.

Confocal laser scanning microscopy Sections of the used ETT will also be analysed using fluorescent in situ hybridization using organism specific Peptide Nucleic Acid (PNA) probes. Each specific probe will be conjugated with a distinct fluorescent label to allow for spatial location and distribution of target organisms (S. aureus, P. aeruginosa, Candida albicans, S. mutans) within the ETT biofilm.

Collection of other data: Baseline demographics of patients will be recorded, including age, sex, APACHE II score, co-morbidities, days from hospital admission, and recent antibiotic administration.

A Zsigmondy and DMFT (decayed, missing, filled teeth) score will be recorded by a dental hygienist during the study to assess the baseline dental status of patients enrolled.

Outcome measures: Primary outcome: Daily plaque and gingival scores following mechanical cleaning, with identification and quantification of bacteria within plaque. Quantitative comparisons will be ascertained from the total log transformed CFU counts and plaque and gingival scores from the two cleaning methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years
* Patients mechanically ventilated with an oral endotracheal tube ->20 teeth with symmetric distribution

Exclusion Criteria:

* Absence of an oral endotracheal tube
* Age <18 years
* <20 teeth or asymmetric distribution
* Expected to be intubated less than 24-hours from recruitment
* Thrombocytopaenia (platelet count <30)
* Uncontrolled coagulopathy
* Suffering from facial or oral trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Modified Silness and Loe plaque and gingival index following cleaning of teeth | Daily until day seven
  The Silness and Loe plaque and gingival index scores plaque and gum disease as 0,1,2, or 3 for each tooth. The index is derived by adding scores and dividing by the number of teeth examined (maximum score 3, minimum 0). The index will be compared between teeth cleaned with a toothbrush versus those cleaned with a swab

SECONDARY OUTCOMES:
Quantitative comparisons of bacterial counts following the two cleaning methods | Daily until day seven

CONTACTS AND LOCATIONS:
Overall Officials: Matt P Wise, DPhil, Principal Investigator — University Hospital of Wales Cardiff & Vale University Health Board
Locations (1):
- Adult Critical Care University Hospital of Wales, Cardiff, South Glamorgan, United Kingdom

REFERENCES:
- [Derived] Marino PJ, Hannigan A, Haywood S, Cole JM, Palmer N, Emanuel C, Kinsella T, Lewis MA, Wise MP, Williams DW. Comparison of foam swabs and toothbrushes as oral hygiene interventions in mechanically ventilated patients: a randomised split mouth study. BMJ Open Respir Res. 2016 Oct 14;3(1):e000150. doi: 10.1136/bmjresp-2016-000150. eCollection 2016. PMID 27843549